CLINICAL TRIAL: NCT01119898
Title: A Phase 2, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Clinical Study to Evaluate the Safety and Efficacy of PENNSAID Gel in the Symptomatic Treatment of Osteoarthritis of the Knee
Brief Title: Exploratory Study of PENNSAID Gel to Treat Symptoms of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COV05100031
Record Dates: First submitted 2010-04-28; First posted 2010-05-10 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Arthritis; NSAIDs; Topical NSAID; Diclofenac; PENNSAID
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PENNSAID Gel (Experimental): Diclofenac sodium 2.0% w/w
  Interventions: Drug: PENNSAID Gel
- Vehicle (Placebo Comparator): The complete carrier containing ingredients at the same concentrations as experimental arm without diclofenac sodium
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: PENNSAID Gel — 2 mL applied to the front, back and sides of the knee twice a day (morning and night) for 4 weeks
  Other Names: diclofenac sodium 2.0% w/w
  Arms: PENNSAID Gel
Drug: Vehicle — 2 mL applied to the front, back and sides of the knee twice a day (morning and night) for 4 weeks
  Arms: Vehicle

SUMMARY:
Osteoarthritis (OA) is the most common form of arthritis. It can cause pain, swelling, and reduced motion in the joints. That can reduce quality of life.

OA can occur in any joint, but usually affects the hands, knees, hips or spine.

The purpose of this study is to find out if doctors might be able to use 2% PENNSAID gel to treat OA in the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Primary osteoarthritis of the knee
2. Radiologic evidence of OA of the knee
3. On stable pain therapy with an oral or topical NSAID or acetaminophen
4. Experience a "moderate flare" of pain following washout of stable pain therapy
5. Able to read and understand English or Spanish to answer pain assessment questions without any explanation
6. If female, surgically sterile or non-pregnant
7. Except for OA, in reasonably good general health
8. Written informed consent

Exclusion Criteria:

1. Secondary OA of the study knee
2. History of pseudo gout or inflammatory flare-ups
3. Participation would conflict with contraindications, warnings or precautions as stated in the prescribing information for oral or topical diclofenac
4. Severe, uncontrolled cardiac, renal, hepatic, or other systemic disease
5. Any malignancy within the previous 3 years, except local therapy for superficial skin cancer not on the study knee
6. Known sensitivity to the use of oral or topical diclofenac, aspirin [acetylsalicylic acid (ASA)] or any other NSAID, dimethyl sulfoxide (DMSO), or ethanol
7. Ongoing abnormality that could confound interpretation of the safety results (eg, anemia, unresponsive gastrointestinal [GI] reflux, etc.)
8. Documented gastroduodenal ulcer or any GI bleeding (except hemorrhoidal) within the last 6 months
9. Uncontrolled diabetes
10. Screening laboratory test results of serum creatinine ≥ 1.5 times upper limit of normal; aspartate aminotransferase (AST), alanine aminotransferase (ALT), or gamma-glutamyltransferase (GGT) ≥ 3 times upper limit of normal; and hemoglobin less than or equal to lower limit of normal
11. Documented alcohol or drug abuse within 1 year
12. If female, breast-feeding
13. Major surgery or previous damage to the study knee at any time, or minor knee surgery to the study knee within 1 year
14. Requires oral or intra-muscular corticosteroids, or received an intra articular corticosteroid injection into the study knee within the past 90 days, or into any other joint within the past 30 days, or currently applying topical corticosteroids onto the study knee
15. Received intra-articular viscosupplementation (eg, hylan G-F 20 [Synvisc®]) in the study knee in the past 6 months
16. On prior stable therapy (ie, more than 3 days per week for the previous month) with an opioid analgesic prior to the screening visit will be excluded.
17. Recently started taking a sedative hypnotic medication for insomnia
18. Taking anti-depressants
19. Not willing to discontinue prohibited medications/therapies
20. Cannot tolerate acetaminophen
21. Re-entering study after dropping out or withdrawn from study
22. Used another investigational drug within the previous 30 days
23. On or currently applying for disability benefits on the basis of knee OA
24. History of fibromyalgia
25. Other painful or disabling conditions affecting the knee or leg, or disabling condition of the hands (used to apply the study drug)
26. Skin disorder with current involvement on the hands (used to apply the study drug) or the knee(s) (application site)
27. Referred to an orthopedic surgeon for consideration of, or been advised to have, knee replacement or knee reconstruction surgery
28. Radiologic evidence of OA of the knee advanced to the point that all cartilage has been eroded (ie, bone on bone)
29. Recently started using a cane within the past 30 days
30. History of chronic headaches that may require more than occasional use of rescue medication for headaches

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2010-08-02 (Actual); Primary Completion 2011-02-16 (Actual); Study Completion 2011-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pierro, MD, Study Director — Mallinckrodt
Locations (26):
- United States (26):
  - Genova Clinical Research, Tucson, Arizona
  - Benchmark Research, Sacramento, California
  - Tampa Bay Medical Research, Inc, Clearwater, Florida
  - Avail Clinical Research, DeLand, Florida
  - Comprehensive NeuroScience Inc., St. Petersburg, Florida
  - Drug Studies America, Marietta, Georgia
  - South Coast Medical Group, Savannah, Georgia
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Sterling Research, Erlanger, Kentucky
  - Radiant Research Inc., St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Clinical Study Center of Asheville, Asheville, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Sterling Research, Cincinnati, Ohio
  - Radiant Research Inc., Columbus, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Radiant Research Inc., Anderson, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Holston Medical Group Clinical Research, Kingsport, Tennessee
  - Benchmark Research, Fort Worth, Texas
  - Benchmark Research, San Angelo, Texas
  - Sun Research Institute, San Antonio, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - HypotheTest, LLC, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wadsworth LT, Kent JD, Holt RJ. Efficacy and safety of diclofenac sodium 2% topical solution for osteoarthritis of the knee: a randomized, double-blind, vehicle-controlled, 4 week study. Curr Med Res Opin. 2016;32(2):241-50. doi: 10.1185/03007995.2015.1113400. Epub 2015 Nov 17. PMID 26506138

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One person who failed screening was randomized in error, but did not receive study drug.
Period: Overall Study
Arm/Group | PENNSAID Gel | Vehicle
Started | 131 | 129
Received Study Drug (mITT) | 130 | 129
Completed | 123 | 117
Not Completed | 8 | 12
Not completed — Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Medical procedure | 1 | 0
Not completed — Randomized in error did not participate | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) - all participants who were randomized and received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | PENNSAID Gel | Vehicle | Total
Number analyzed (Participants) | 130 | 129 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.23) | 61.9 (9.07) | 61.1 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 90 | 174
  Male | 46 | 39 | 85
Region of Enrollment [Number; unit: participants]
  United States | 130 | 129 | 259

OUTCOME MEASURES:

1. Primary Outcome: Pain When Walking On A Flat Surface
Description: Participants rate their pain intensity when walking on a flat surface as none, mild, moderate, severe or extreme. The number of participants who rate their pain in each category is presented.
Time Frame: at Baseline
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 130 | 129
Participants
  None | 0 | 1
  Mild | 8 | 4
  Moderate | 62 | 67
  Severe | 51 | 43
  Extreme | 9 | 14

2. Primary Outcome: Pain When Walking On A Flat Surface
Description: as for outcome 1
Time Frame: at Week 4
Population: mITT population with non-missing data at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 123 | 118
Participants
  None | 19 | 19
  Mild | 47 | 38
  Moderate | 45 | 51
  Severe | 11 | 10
  Extreme | 1 | 0

3. Primary Outcome: Pain When Going Up Or Down Stairs
Description: Participants rate their pain intensity when going up or down stairs as none, mild, moderate, severe or extreme. The number of participants who rate their pain in each category is presented.
Time Frame: at Baseline
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 130 | 129
Participants
  None | 0 | 0
  Mild | 1 | 1
  Moderate | 14 | 14
  Severe | 80 | 84
  Extreme | 35 | 30

4. Primary Outcome: Pain When Going Up Or Down Stairs
Description: as for outcome 3
Time Frame: at Week 4
Population: mITT population with non-missing data at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 123 | 118
Participants
  None | 4 | 4
  Mild | 34 | 32
  Moderate | 51 | 37
  Severe | 29 | 40
  Extreme | 5 | 5

5. Primary Outcome: Pain At Night While In Bed
Description: Participants rate their pain intensity at night while in bed as none, mild, moderate, severe or extreme. The number of participants who rate their pain in each category is presented.
Time Frame: at Baseline
Population: mITT population with non-missing data at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 129 | 129
Participants
  None | 5 | 6
  Mild | 23 | 26
  Moderate | 60 | 50
  Severe | 32 | 33
  Extreme | 9 | 14

6. Primary Outcome: Pain At Night While In Bed
Description: as for outcome 5
Time Frame: at Week 4
Population: mITT population with non-missing data at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 123 | 118
Participants
  None | 37 | 30
  Mild | 45 | 45
  Moderate | 34 | 35
  Severe | 5 | 8
  Extreme | 2 | 0

7. Primary Outcome: Pain While Sitting Or Lying Down
Description: Participants rate their pain intensity while sitting or lying down as none, mild, moderate, severe or extreme. The number of participants who rate their pain in each category is presented.
Time Frame: at Baseline
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 130 | 129
Participants
  None | 1 | 4
  Mild | 30 | 22
  Moderate | 63 | 63
  Severe | 30 | 28
  Extreme | 6 | 12

8. Primary Outcome: Pain While Sitting Or Lying Down
Description: as for outcome 7
Time Frame: at Week 4
Population: mITT population with non-missing data at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 123 | 118
Participants
  None | 36 | 25
  Mild | 46 | 55
  Moderate | 36 | 34
  Severe | 5 | 4
  Extreme | 0 | 0

9. Primary Outcome: Pain While Standing
Description: Participants rate their pain intensity while standing as none, mild, moderate, severe or extreme. The number of participants who rate their pain in each category is presented.
Time Frame: at Baseline
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 130 | 129
Participants
  None | 0 | 2
  Mild | 7 | 6
  Moderate | 54 | 52
  Severe | 53 | 51
  Extreme | 16 | 18

10. Primary Outcome: Pain While Standing
Description: as for outcome 9
Time Frame: at Week 4
Population: mITT population with non-missing data at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | PENNSAID Gel | Vehicle
Number analyzed (Participants) | 123 | 118
Participants
  None | 15 | 13
  Mild | 47 | 42
  Moderate | 49 | 50
  Severe | 11 | 11
  Extreme | 1 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were only counted once for each body system/preferred term.
Arm/Group | PENNSAID Gel | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/129
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/129
Other Adverse Events (participants affected / at risk) | 45/130 | 59/129
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PENNSAID Gel (N=130) | Vehicle (N=129)
Application site dryness (General disorders) | 28 | 28
Application site exfoliation (General disorders) | 9 | 11
Application site erythema (General disorders) | 5 | 15
Application site pruritis (General disorders) | 3 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes